CLINICAL TRIAL: NCT05638633
Title: Prednisolone and Vitamin B1, B6, and B12 in Patients With Post-COVID-19-Syndrome (PC19S) - a Randomized Controlled Trial in Primary Care
Brief Title: Prednisolone and Vitamin B1/6/12 in Patients With Post-Covid-Syndrome
Acronym: PreVitaCOV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University Hospital Tuebingen (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F001AM02222_1; 2022-001041-20 (EudraCT Number)
Record Dates: First submitted 2022-11-18; First posted 2022-12-06 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Post-COVID-19 Syndrome
Keywords: Prednisolone; Vitamin B1; Vitamin B6; Vitamin B12; PC19S; Fatigue; ME/CFS (myalgic encephalomyelitis/chronic fatigue syndrome)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue; Fatigue Syndrome, Chronic | interventions — Prednisolone; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: after Baseline, Randomization to 4 arms:
  1. st arm (prednisolone and placebo)
  2. nd arm (placebo an Vitamin B compound)
  3. rd arm (prednisolone and Vitamin B compound)
  4. th arm (placebo and placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: blinded labelling of the study drug by the Hospital pharmacy of the Charité
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1st arm (prednisolone and placebo) (Active Comparator): Day 1-5: prednisolone 20mg 1x1 and placebo 1x1 Day 6-28: prednisolone 5mg 1x1 and placebo 1x1
  Interventions: Drug: Prednisolone 20 mg/ 5 mg; Drug: Placebo for Vitamin B compound
- 2nd arm (placebo and Vitamin B compound) (Active Comparator): Day 1-5: Placebo 1x1 and Vitamin B compound (100 mg B1, 50 mg B6, 500µ B12) 1x1 Day 6-28: placebo 1x1 and Vitamin B compound (100 mg B1, 50 mg B6, 500 µg B12) 1x1
  Interventions: Drug: Vitamin B compound (100mg B1, 50 mg B6, 500 µg B12); Drug: Placebo for Prednisolon
- 3rd arm (prednisolone and Vitamin B compound) (Active Comparator): Day 1-5: prednisolone 20mg 1x1 and Vitamin B compound (100 mg B1, 50 mg B6, 500µg B12) 1x1 Day 6-28: prednisolone 5mg 1x1 and Vitamin B compound (100 mg B1, 50mg B6, 500µg B12) 1x1
  Interventions: Drug: Prednisolone 20 mg/ 5 mg; Drug: Vitamin B compound (100mg B1, 50 mg B6, 500 µg B12)
- 4rd arm (placebo and placebo) (Placebo Comparator): Day 1-5: Placebo 1x1 and placebo 1x1 Day 6-28: placebo 1x1 and placebo 1x1
  Interventions: Drug: Placebo for Vitamin B compound; Drug: Placebo for Prednisolon

INTERVENTIONS:
Drug: Prednisolone 20 mg/ 5 mg — Administration of prednisolone 20 mg for 5 days, followed by prednisolone 5 mg for 23 days.
  Other Names: N.I.
  Arms: 1st arm (prednisolone and placebo); 3rd arm (prednisolone and Vitamin B compound)
Drug: Vitamin B compound (100mg B1, 50 mg B6, 500 µg B12) — Administration of vitamin B compound for 28 days.
  Other Names: Vitamin B complex forte
  Arms: 2nd arm (placebo and Vitamin B compound); 3rd arm (prednisolone and Vitamin B compound)
Drug: Placebo for Vitamin B compound — Administration of placebo for vitamin B compound placebo for 28 days.
  Other Names: N.I.
  Arms: 1st arm (prednisolone and placebo); 4rd arm (placebo and placebo)
Drug: Placebo for Prednisolon — Administration of placebo for prednisolone 20 mg for 5 days, followed by placebo for prednisolone 5 mg for 23 days.
  Other Names: N.I.
  Arms: 2nd arm (placebo and Vitamin B compound); 4rd arm (placebo and placebo)

SUMMARY:
This is a multicenter, randomized, placebo controlled, double-blind phase III trial with four parallel groups studying studying the feasibility of RCT in primary care as well as the effectiveness of treatment with prednisolone and/or vitamin B1/6/12 for PC19S.

DETAILED DESCRIPTION:
PC19S affects a considerable portion of patients after an infection with SARS-CoV-2 with a broad range of disabling symptoms. Neurotropic vitamins such as vitamins B1, B6, an B12, and drugs with anti-inflammatory properties such as corticosteroids were suggested to alleviate symptoms. The trial is designed as a two-step approach that will

1. prove the feasibility of recruitment and retention of patients with PC19S in a primary care setting (pilot study, n=100)
2. investigate the effectiveness and safety of the treatment drugs alone and of their combination (confirmatory study, n= 340).

The pilot study will be transformed into a confirmatory study if feasibility is given, defined as retention rate of 85% after enrollment of 100 patients. Or on recommendation of the Data Safety and Monitoring Board (DSMB).

In addition, blood samples wil be analysed for routine parameters and vitamin B12 derivates as well as cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (at least 18 years old)
2. history of SARS-CoV-2 infection at least 12 weeks ago (the infection must be documented by either a positive PCR or antibody-Test or be confirmed by the patient's GP)
3. symptoms concerning at least one of the following domains: fatigue, dyspnea, cognition, anxiety, depression
4. above mentioned symptom(s) that developed during or after the SARS-CoV-2 infection, that persist until study inclusion, and that are associated with COVID 19 as assessed by the patients' general practitioner or the local investigator

Exclusion Criteria:

1. acute Coronavirus disease (COVID-19) at baseline visit
2. patients who were treated in the intensive care unit because of COVID-19
3. pregnancy/ breastfeeding
4. diabetes mellitus
5. PC19S symptoms that can be explained by an alternative diagnosis
6. History of severe medical conditions such as

   * concomitant acute infectious disease
   * gastrointestinal ulcer
   * liver disease/liver cirrhosis
   * malabsorption or condition after bariatric surgery
   * chronic airway disease
   * chronic heart failure [New York Heart Association (NYHA) III and IV]
   * neurological disorders
   * untreated hypothyroidism
   * significantly impaired glucuronidation
   * immunodeficiency or a chronically weakened immune system
   * mental disorders
   * active cancer
   * any other severe medical conditions that preclude participation as determined by responsible physician
7. current use of

   * immunosuppressive drugs
   * non-steroidal antiinflammatory drugs (NSAID)
   * fluoroquinolones
   * anticoagulation
   * any other drug that could exhibit clinically relevant interactions with the study medication (as described in Fachinformation Prednisolon STADA®, Predni H Tablinen® Zentiva or Fachinformation Vitamin B komplex Hevert). The decision on the clinical relevance of the interactions is at the discretion of the clinical investigator.
8. systemic treatment with prednisolone for at least 7 days or any parenteral application since the end of the acute phase of COVID-19; treatment with vitamins B1, B6, or B12 in doses equivalent to the dose of the study medi-cation for at least 7 days or any parenteral application since the end of the acute phase of COVID-19; vitamin supplements containing vitamin B1, B6, or B12 should have been ceased at least 4 weeks prior to the inclusion of the study
9. known allergies and contraindications to the intervention drugs
10. need of care and/or peer dependency
11. nursing home residents
12. inability to understand the scope of the study, to follow study procedures and to give informed consent or to attend the study sites
13. participation in another interventional trial at the same time or within the past 3 months before enrolment
14. female patients considering to get pregnant during the first month of the trial and within 1 week after the last dose of study drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Pilot phase: Proportion of participants retained after 28 days | 4 weeks
  feasibility and acceptance of screening and recruitment in primary care; aim > 85 % retention rate of 100 patients enrolled
Confirmatory phase: Mean difference in PROMIS Total Score from day 0 to day 28 | 4 weeks
  change in symptom severity to day 28 as assessed by specifically tailored total score based on the patient reported outcome measurement information system (PROMIS)

SECONDARY OUTCOMES:
PROMIS total and subscores | 6 months
  Severity of each PC19 symptom domain (patient reported outcome measurement information system (PROMIS))
Measure Yourself Medical Outcome Profile (MYMOP) | 6 months
  Severity of three subjectively chosen PC19 symptoms
Overall assessment of functional status | 6 months
  Severity of PC19 symptom burden
PC19 symptom list | 6 months
  checklist, number of subjectively present symptoms
EQ-5D-5L | 6 months
  Health related quality of life, 5 point rating scale, 0 to 20 points, higher scores indicate worse outcomes
visual analogue scale | 6 months
  Health related quality of life, 0 to 100 points, higher scores indicate a better outcome
PHQ 8 | 6 months
  Depression, 4 point rating scale, 0 to 24 points possible, higher scores indicate a worse outcome
Chalder Scale | 6 months
  Fatigue, 4 point rating scale, 0 to 33 points possible, higher values indicate a worse outcome
Numeric rating scale for pain | 6 months
  Pain, 10 point rating scale, higher values indicate a worse outcome
Testbatterie zur Aufmerksamkeitsprüfung (TAP) | 4 weeks
  cognitive function (Alertness: reaction time, distractibility: omissions and reaction time, divided attention: omissions, visual scanning: omissions and reaction time, flexibility: reaction time and errors)
Physical exercise | 6 months
  1minute Sit-to-Stand-Test, number of repetitions, BORG Scale, oxygen-saturation
Use of on-demand medication and change in concomitant medication | 6 months
  intake of on-demand medication, daily drug doses
qualitative assessment of acceptance | 6 months
  qualitative interviews with subgroup sample
feasibility/acceptance | 6 months
  exploratory questionnaire, rating scales and grades

CONTACTS AND LOCATIONS:
Overall Officials: Ildikó Gágyor, Prof. Dr., Study Director — Director of Institute for General Practice Würzburg University Hospital
Locations (3):
- Germany (3):
  - University Hospital Wuerzburg, Würzburg, Bavaria
  - Unversity Hospital Schleswig-Holstein, Kiel
  - University Hospital Tuebingen, Tübingen

IPD SHARING:
Plan to Share IPD: No